CLINICAL TRIAL: NCT02755792
Title: Can Chinese Calligraphy Writing Enhance Cognitive Performance and Emotional Calmness in Older Adults With Mild Cognitive Impairment? A RCT Study
Brief Title: Calligraphy Writing for Cognitive and Emotional Enhancement Among Older MCI People
Acronym: CALLI-MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Prof. Chetwyn Chan, Associate Vice President (Learning and Teaching) and Chair Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Calligraphy-MCI
Record Dates: First submitted 2016-04-22; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognitive training; Calligraphy; Emotional calmness; Working memory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calligraphy Training (Experimental): This group receives a Chinese calligraphy training program of 16 sessions over 8 weeks in a class of 8-12 participants. Each session is 1.5 hours.
  Interventions: Behavioral: Calligraphy Training
- iPad Training (Active Comparator): This group receives an iPad training program of 16 sessions over 8 weeks in a class of 8-12 participants. Each session is 1.5 hours.
  Interventions: Behavioral: iPad Training

INTERVENTIONS:
Behavioral: Calligraphy Training
  Arms: Calligraphy Training
Behavioral: iPad Training
  Arms: iPad Training

SUMMARY:
This study is aimed to investigate the efficacy of an 12-week Chinese calligraphy training program for enhancing cognitive and emotional functions of older adults with mild cognitive impairment. Participants are tested with several cognitive tests and electroencephalography (EEG), psycho-physical parameters and brain activities are recorded. Results are compared at pre-intervention, post-intervention, and 6-month post-intervention to provide evidence of benefits of Chinese calligraphy practice.

DETAILED DESCRIPTION:
Participants are older adults with mild cognitive impairment, who will be recruited from several community elderly centers in Hong Kong according to selective criteria. The participants are randomly assigned to an experimental or a control group. The experimental group is invited to participate in 16 sessions of structured Chinese calligraphy program over 12 weeks. Each session lasts for 1.5 hours. The control group is invited to participate in an iPad learning program with navigating the Internet. The iPad program is also consisted of 16 sessions of 1.5 hours each over 8 weeks. Cognitive tests and physiological measures are conducted immediately before and after intervention and at 6-month post-intervention follow-up. Statistical analysis are performed to investigate the significant differences and interactions among the three time points. The association of cognitive performance and emotional calmness is also investigated.

Selected participants are invited to take part in a EEG session while doing some computer tasks related to Chinese calligraphy. EEG results of are used to explore neural activities associated with visuospatial working memory and to provide evidence for neural changes at functional level as a result of Chinese calligraphy training and practice.

ELIGIBILITY:
Inclusion Criteria:

* Meeting Petersen's criteria for mild cognitive impairment
* Being able to read simple Chinese characters
* Community-dwelling
* Clinical Dementia Rating score of 0.5
* No substantial prior experience of calligraphy writing
* Willing to write using a brush and willing to participate

Exclusion Criteria:

* Presence of musculoskeletal problems preventing participants from writing
* Known chronic cardiovascular (e.g. systolic BP > 140mmHg) or pulmonary conditions requiring long-term medication
* Presence of severe mental disorder such as psychosis or depression.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Digit span backward test (DSB) from baseline, after end of training, and 6-month follow-up. | Baseline, within 2 weeks after end of training, and 6-month follow-up.
  DSB evaluates working memory, which requires recalling digits in reverse order. The DSB test is structured with increased levels of difficulty.

SECONDARY OUTCOMES:
Color Trails Test (CTT) | Baseline, within 2 weeks after end of training, and 6-month follow-up.
  CTT is consisted of two parts. CTT 1 evaluates attention and perceptual speed. Participants are asked to draw a line to between circles in consecutive order numbered 1 - 25, as quickly as possible. CTT 2 evaluates set-shifting. Each number (1 - 25) of CTT 2 is printed twice, one in pink and another in yellow color circle. Subjects are asked to connect the numbers in consecutive order but alternating between pink and yellow.
Symbol-digit Modalities Test (SDMT) | Baseline, within 2 weeks after end of training, and 6-month follow-up.
  SDMT evaluates executive function, in particular mental flexibility, of older people with cognitive impairment. It is a simple substitution task in which participants are asked to substitute series of symbols with specific digits within a period of 90 seconds.
Heart rate and heart rate variability. | At the week 1, 5, 9, 12 during the intervention period, and at 6-month post-intervention.
  It is measured by the Polar RS800C.
Blood pressure. | At the week 1, 5, 9, 12 during the intervention period, and at 6-month post-intervention.
  It is measured by the Portapres.
Geriatric Depression Scale - Short Form (GDS-SF) | Baseline, within 2 weeks after end of training, and 6-month post-intervention.
  GDS-SF measures subjective appraisal of the mood state. It consists of 15 statements about various aspects of mood such as appetite, quality of sleep, hope, and social functioning. Each statement is responded using a dichotomous format (yes/no).
Consortium to Establish a Registry for Alzheimer's Disease - Neuropsychological Assessment Battery (CERAD-NAB) | Baseline, within 2 weeks after end of training, and 6-month post-intervention.
  CERAD-NAB is used to ask subjects to recall or identify the list of words learnt after a five minute delay.

CONTACTS AND LOCATIONS:
Overall Officials: Chetwyn CH Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

REFERENCES:
- [Background] Gauthier S, Reisberg B, Zaudig M, Petersen RC, Ritchie K, Broich K, Belleville S, Brodaty H, Bennett D, Chertkow H, Cummings JL, de Leon M, Feldman H, Ganguli M, Hampel H, Scheltens P, Tierney MC, Whitehouse P, Winblad B; International Psychogeriatric Association Expert Conference on mild cognitive impairment. Mild cognitive impairment. Lancet. 2006 Apr 15;367(9518):1262-70. doi: 10.1016/S0140-6736(06)68542-5. PMID 16631882
- [Background] Belleville S, Chertkow H, Gauthier S. Working memory and control of attention in persons with Alzheimer's disease and mild cognitive impairment. Neuropsychology. 2007 Jul;21(4):458-69. doi: 10.1037/0894-4105.21.4.458. PMID 17605579
- [Background] Boyle PA, Malloy PF, Salloway S, Cahn-Weiner DA, Cohen R, Cummings JL. Executive dysfunction and apathy predict functional impairment in Alzheimer disease. Am J Geriatr Psychiatry. 2003 Mar-Apr;11(2):214-21. PMID 12611751
- [Background] Chan WC, Lam LC, Tam CW, Lui VW, Chan SS, Chan WM, Chiu HF. Prevalence of neuropsychiatric symptoms in chinese older persons with mild cognitive impairment-a population-based study. Am J Geriatr Psychiatry. 2010 Oct;18(10):948-54. doi: 10.1097/JGP.0b013e3181d69467. PMID 20808089
- [Background] Wilson RS, Scherr PA, Schneider JA, Tang Y, Bennett DA. Relation of cognitive activity to risk of developing Alzheimer disease. Neurology. 2007 Nov 13;69(20):1911-20. doi: 10.1212/01.wnl.0000271087.67782.cb. Epub 2007 Jun 27. PMID 17596582
- [Background] Belleville S, Gilbert B, Fontaine F, Gagnon L, Menard E, Gauthier S. Improvement of episodic memory in persons with mild cognitive impairment and healthy older adults: evidence from a cognitive intervention program. Dement Geriatr Cogn Disord. 2006;22(5-6):486-99. doi: 10.1159/000096316. Epub 2006 Oct 16. PMID 17050952